CLINICAL TRIAL: NCT03267004
Title: Validation Study of a Passive Image-Assisted Dietary Assessment With Automated Image Analysis Process
Brief Title: Dietary Assessment Study Via Digital Images
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Faculty Advisor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: UTK IRB-17-03829-XP
Record Dates: First submitted 2017-08-10; First posted 2017-08-30 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Diet Habit
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: A 2x2x2x2x3 mixed factorial design will be used, with a between-subject factor of the order of meals (Order 1 and 2) and within-subject factors of food shapes (Regular and Irregular), food complexities (Single food and Mixed food), meals (Meal A and B), and methods of measurement (DietCam, weighed food intake, and 24-hour dietary recall).
Who Masked: Investigator
Masking Description: The project staffs who will be analyzing the digital images taken by Sony Smarteyeglass during meal sessions will be masked including the types of foods and volume provided to the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Meal Order 1 (Experimental): Meal A will be served to participant in meal session 1 and Meal B in meal session 2.
  Interventions: Device: Dietary Assessment of Meal A using images taken by Sony Smarteyeglass; Device: Dietary Assessment of Meal B using Images taken by Sony Smarteyeglass
- Meal Order 2 (Experimental): Meal B will be served to participant in meal session 1 and Meal A in meal session 2.
  Interventions: Device: Dietary Assessment of Meal A using images taken by Sony Smarteyeglass; Device: Dietary Assessment of Meal B using Images taken by Sony Smarteyeglass

INTERVENTIONS:
Device: Dietary Assessment of Meal A using images taken by Sony Smarteyeglass — Participant will be wearing Sony Smarteyeglass to record digital images while eating meal A in the laboratory
  Meal A:
  Turkey and Provolone Cheese Sandwich [whole wheat bread 52g(female & male), Turkey 70g(female) & 133g(male), Provolone cheese 23g(female & male), tomato 50g(female & male), lettuce 45g(female & male)]; Chicken and wild rice [chicken 98g(female & male), wild rice 71g(female) & 107g(male)]; chocolate chips cookies [44g(female) & 60.5g(male)]; potato chips [39g(female) & 52g(male)].
Device: Dietary Assessment of Meal B using Images taken by Sony Smarteyeglass — Participant will be wearing Sony Smarteyeglass to record digital images while eating meal B in the laboratory
  Meal B:
  Ham & Cheddar cheese wrap [Tortilla 45g(female & male), Ham deli 76g(female) & 103g(male), cheddar cheese 21g(female) & 32g(male), Spring Mix 36g(female & male), Fat Free ranch dressing 29g(female & male)]; Pasta with broccoli and Alfredo sauce [Pasta 91g(female) & 121g(male), Broccoli 66g(female & male), Alfredo sauce 38g(female) & 50g(male)]; Chocolate Ice-cream [107g(female), 138g(male)]; Red seedless grapes [365g (female), 471g(male)].

SUMMARY:
The purpose of this investigation is to validate a passive image-assisted dietary assessment method using images taken by Sony Smarteyeglass and an automatic image analysis software, DietCam, to identify food items and estimate portion sizes. Participants will be randomized into one of the two orders of meals (Order 1 and 2). In each meal, participants will be given a meal that includes a regular-shaped single food (i.e., cookie), an irregular-shape single food (i.e., ice cream), a regular-shaped mixed food (i.e., sandwich), and irregular-shaped mixed food (i.e., pasta dish).

DETAILED DESCRIPTION:
All participants will be asked to come to Healthy Eating and Activity Laboratory for 1, 30-minute screening session, and then for 2, 40-minute meal sessions, with approximately one week occurring between each session. Sessions will be scheduled between 11:00am and 5:00pm, Monday to Friday. During the screening session, interested participants will sign the consent form. After signing the consent from, eligibility will be confirmed by taking height and weight measures. Participants will also be given questionnaires related to demographics. Prior to the start of the first meal session, eligible participants will be randomized to one of the two orders (Order 1 and 2), using a random numbers table. Participants will be instructed for the meal sessions to stop eating a minimum of two hours prior to the scheduled meal sessions and only consume water during that period.

During both meal sessions, instructions on how to use Sony Smarteyeglass will be provided to participants. These instructions will include how to wear and use the eyeglasses. Participants will be instructed that, after putting on the Smarteyeglass, to initiate the recording via the controller of the Sony Smarteyeglass. After the recording is initiated and prior to starting to eat, participants will be instructed to look at each provided food at the table. Then, participants will also be instructed to turn their head toward the left shoulder, look at each food from the side, and then repeat the same step for turning their head toward the right shoulder. Participants will be asked to start the meal by taking one bite of each provided food. For the first bite of each food, participants will be instructed to hold the food, either in their hand or on a fork or spoon (depending on the food), approximately 12 inches in front of the eyeglasses and to look at the food. Following taking the first bite of each provided food, participants will be instructed to eat normally until satisfied. Participants will be given 30 minutes to eat. The investigator will leave the room while the participant is eating. The investigator will check in with participants every 10 minutes. At the end of 30 minutes, participants will be instructed to again look at each provided food on the table at three different angles (looking straight at each food, from left side and the right side) following the exact same procedure at the beginning of the meal.

On the day following each meal session, participants will be called to complete a 24-hour dietary recall, which will take 20 minutes to complete. Instructions will be provided to participants at the end of each meal session about how to complete the dietary recall and a two-dimensional visual aid will be provided to aid participants in estimating the consumed portions for each food and beverage item consumed.

The second meal session will follow the same procedure as the first session. At the end of second meal session, participants will be asked to complete a questionnaire to provide feedback on their use of the Sony Smarteyeglass.

For the first and second meal session, the meals will contain foods that are categorized into two food shapes (Regular and Irregular) and two food complexities (Single food and Mixed food). Each meal will contain four foods with the four foods representing the four potential food categories (regular-shaped single food, irregular-shaped single food, regular-shaped mixed food, irregular-shaped mixed food). Along with the four foods, participants will be given 20oz of water in each meal session. Foods will be weighed prior to being provided to participants and the amount provided to participants will be within +/- 3g of the amount calculated. Mixed foods will be broken down into their individual food components and measured. Each meal will provide approximately 50% of daily estimated energy need for each sex. The Estimated Calories Needed Per Day for males and females aged 19 to 35 years are 2450 kcal/day and 1900 kcal/day, respectively. Thus, each meal will provide approximately 1225 kcal for males and 950 kcal for females. Each food will provide approximately 25% of the energy for each meal.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 65 years;
* body mass index (BMI) 18.5 to 24.9 kg/m2;
* no food allergies/intolerance to foods used in the investigation;
* report not having a dietary plan or dietary restrictions that prevents consumption of the foods used in the investigation;
* report a favorable preference for the foods served in the meal, with participants rate each food item 3 on a Likert scale during the phone screen;
* able to complete all two meal sessions within four weeks of the screening session;
* are not legally blind without corrected lenses; and
* are able to eat a meal while wearing the Sony Smarteyeglass.

Exclusion Criteria:

* wear electronic medical devices such as pacemakers and implantable defibrillators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2020-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsz-Kiu Chui, Principal Investigator — University of Tennessee
Locations (1):
- Healthy Eating and Activity Laboratory, University of Tennessee, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] U.S. Department of Health and Human Services; U.S. Department of Agriculture. 2015-2020 Dietary guidelines for Americans. Appendix 2. Estimated Calorie Needs per Day, by Age, Sex, and Physical Activity Level 2015; 8th Edition:http://health.gov.dietaryguidelines/2015/guidelines/. Accessed April 18, 2017.
- [Background] Lohman TR, Roche AF, Martorell R. Anthropometric Standardization Reference Manual. Champaign,Illinois: Human Kinetics Books; 1988.
- [Background] He H, Kong F, Tan J. DietCam: Multiview Food Recognition Using a Multikernel SVM. IEEE J Biomed Health Inform. 2016 May;20(3):848-855. doi: 10.1109/JBHI.2015.2419251. Epub 2015 Apr 2. PMID 25850095
- [Background] Sony Coporation. Smarteyeglass: API Overview. 2017; https://developer.sony.com/develop/wearables/smarteyeglass-sdk/api-overview/. Accessed Feb, 2017.
- [Derived] Chui TK, Tan J, Li Y, Raynor HA. Validating an automated image identification process of a passive image-assisted dietary assessment method: proof of concept. Public Health Nutr. 2020 Oct;23(15):2700-2710. doi: 10.1017/S1368980020000816. Epub 2020 Jun 10. PMID 32517834

RESULTS

PARTICIPANT FLOW:
Groups:
- Meal Order 1: Meal A will be served to participant in meal session 1 and Meal B in meal session 2.
  Dietary Assessment of Meal A using images taken by Sony Smarteyeglass: Participant will be wearing Sony Smarteyeglass to record digital images while eating meal A in the laboratory
  Meal A:
  Turkey and Provolone Cheese Sandwich [whole wheat bread 52g(female & male), Turkey 70g(female) & 133g(male), Provolone cheese 23g(female & male), tomato 50g(female & male), lettuce 45g(female & male)]; Chicken and wild rice [chicken 98g(female & male), wild rice 71g(female) & 107g(male)]; chocolate chips cookies [44g(female) & 60.5g(male)]; potato chips [39g(female) & 52g(male)].
  Dietary Assessment of Meal B using Images taken by Sony Smarteyeglass: Participant will be wearing Sony Smarteyeglass to record digital images while eating meal B in the laboratory
  Meal B:
  Ham & Cheddar cheese wrap [Tortilla 45g(female & male), Ham deli 76g(female) & 103g(male), cheddar cheese 21g(female) & 32g(male), Spring Mix 36g(female & male), Fat Free ranch dressing 29g(female & male)]; Pasta with broccoli and Alfredo sauce [Pasta 91g(female) & 121g(male), Broccoli 66g(female & male), Alfredo sauce 38g(female) & 50g(male)]; Chocolate Ice-cream [107g(female), 138g(male)]; Red seedless grapes [365g (female), 471g(male)].
- Meal Order 2: Meal B will be served to participant in meal session 1 and Meal A in meal session 2.
  Dietary Assessment of Meal A using images taken by Sony Smarteyeglass: Participant will be wearing Sony Smarteyeglass to record digital images while eating meal A in the laboratory
  Meal A:
  Turkey and Provolone Cheese Sandwich [whole wheat bread 52g(female & male), Turkey 70g(female) & 133g(male), Provolone cheese 23g(female & male), tomato 50g(female & male), lettuce 45g(female & male)]; Chicken and wild rice [chicken 98g(female & male), wild rice 71g(female) & 107g(male)]; chocolate chips cookies [44g(female) & 60.5g(male)]; potato chips [39g(female) & 52g(male)].
  Dietary Assessment of Meal B using Images taken by Sony Smarteyeglass: Participant will be wearing Sony Smarteyeglass to record digital images while eating meal B in the laboratory
  Meal B:
  Ham & Cheddar cheese wrap [Tortilla 45g(female & male), Ham deli 76g(female) & 103g(male), cheddar cheese 21g(female) & 32g(male), Spring Mix 36g(female & male), Fat Free ranch dressing 29g(female & male)]; Pasta with broccoli and Alfredo sauce [Pasta 91g(female) & 121g(male), Broccoli 66g(female & male), Alfredo sauce 38g(female) & 50g(male)]; Chocolate Ice-cream [107g(female), 138g(male)]; Red seedless grapes [365g (female), 471g(male)].
Period: Overall Study
Arm/Group | Meal Order 1 | Meal Order 2
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Meal Order 1 | Meal Order 2 | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (6.2) | 24.8 (7.1) | 25.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants] — nominal scale
  Participants
    Female | 7 | 10 | 17
    Male | 8 | 5 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 12 | 2 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 11 | 14
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Weighed Food Intake
Description: Before and after each meal session, each food items will be weighed to the nearest tenth of a gram using an electronic food scale. Assessing the weight change of food intake.
Time Frame: Meal session 1 and 2 within 4 weeks of initial screening session
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Meal Order 1 | Meal Order 2
Number analyzed (Participants) | 15 | 15
grams | 354.4 (126.2) | 354.4 (126.2)

2. Primary Outcome: 24-hour Dietary Recall
Description: On the following day of each meal session, the investigator will ask the participant to recall their dietary intake by having the participant reporting all foods and beverages consumed and the time in which they consumed these items within the past 24 hours. Participants will be asked what time of day the foods and beverages were consumed and will be shown two-dimensional food shapes to help with estimating portion sizes. Only dietary intake for the meal session will be entered into NDS-R to convert to commonly used measurements.
Time Frame: The following day of meal session 1 and 2 within 4 weeks of initial screening session
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Meal Order 1 | Meal Order 2
Number analyzed (Participants) | 15 | 15
grams | 302.6 (132.6) | 302.6 (132.6)

ADVERSE EVENTS:
Time Frame: 4 weeks of participation
Arm/Group | Meal Order 1 | Meal Order 2
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-05-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT03267004/Prot_002.pdf
  • Informed Consent Form (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT03267004/ICF_001.pdf